CLINICAL TRIAL: NCT00005369
Title: Coronary Artery Disease Mechanisms in High Risk Families--Racial Difference
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4260; R01HL049762 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To examine whether differences existed between asymptomatic white and African Americans known to be at high risk for premature coronary artery disease (CAD) in risk factor distributions, prevalence of occult coronary disease, and mechanisms of coronary disease expression.

DETAILED DESCRIPTION:
BACKGROUND:

The investigators hypothesized that increased platelet activation and coronary artery vasoconstriction exist in African Americans, due to greater vascular endothelial dysfunction, heightened adrenergic drive, and greater vascular reactivity, resulting in excess sudden death and the occurrence of myocardial infarction in people with less severe angiographic coronary disease.

The study was one of eight grants awarded as part of the Request for Applications "Mechanisms Underlying Coronary Heart Disease in Blacks". The initiative was released in October 1991 and awarded in September 1992.

DESIGN NARRATIVE:

Previous studies had demonstrated high prevalences of coronary disease risk factors and occult coronary disease in this sibling population. Subjects were recruited to come for a one day screening, with measurement of coronary disease risk factors (blood pressure, smoking, lipid profile, apolipoproteins B and A1, lipoprotein(a), blood glucose, insulin, and fibrinogen), and a maximal treadmill test with tomographic thallium imaging to identify occult coronary disease. Platelet function was assessed by spontaneous in-vitro aggregation, activated IIa/IIIb receptor density, and serum thromboxane B2 concentration. Factors contributing to sudden cardiac death were assessed by an echocardiogram for left ventricular mass, electrocardiogram (ECG) for QRS late potentials, and 24 hour ECG monitoring for ventricular arrhythmias, episodes of silent ischemia, and heart rate variability (to assess adrenergic drive). Vascular reactivity was characterized by heart rate and blood pressure changes during Stroop color card and cold pressor testing. Siblings with an abnormal exercise ECG and/or thallium scan were offered coronary arteriography to assess the severity of angiographic coronary disease and the vasomotor responses to isometric handgrip and intracoronary acetylcholine, an endothelium-dependent vasodilator. In coronary arteries with minimal angiographic disease, changes in coronary vascular resistance during handgrip and acetylcholine were also measured with a doppler flow velocity catheter and the proximal arteries were imaged with intravascular ultrasound.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1996-08 (Actual)

REFERENCES:
- [Background] Kral BG, Becker LC, Blumenthal RS, Aversano T, Fleisher LA, Yook RM, Becker DM. Exaggerated reactivity to mental stress is associated with exercise-induced myocardial ischemia in an asymptomatic high-risk population. Circulation. 1997 Dec 16;96(12):4246-53. doi: 10.1161/01.cir.96.12.4246. PMID 9416889
- [Background] Allen JK, Young DR, Blumenthal RS, Moy TF, Yanek LR, Wilder L, Becker LC, Becker DM. Prevalence of hypercholesterolemia among siblings of persons with premature coronary heart disease. Application of the Second Adult Treatment Panel guidelines. Arch Intern Med. 1996 Aug 12-26;156(15):1654-60. PMID 8694663
- [Background] Weiss EJ, Bray PF, Tayback M, Schulman SP, Kickler TS, Becker LC, Weiss JL, Gerstenblith G, Goldschmidt-Clermont PJ. A polymorphism of a platelet glycoprotein receptor as an inherited risk factor for coronary thrombosis. N Engl J Med. 1996 Apr 25;334(17):1090-4. doi: 10.1056/NEJM199604253341703. PMID 8598867
- [Background] Blumenthal RS, Becker DM, Moy TF, Coresh J, Wilder LB, Becker LC. Exercise thallium tomography predicts future clinically manifest coronary heart disease in a high-risk asymptomatic population. Circulation. 1996 Mar 1;93(5):915-23. doi: 10.1161/01.cir.93.5.915. PMID 8598082